CLINICAL TRIAL: NCT07123155
Title: A Phase 2, Multicenter, Randomized, Placebo-controlled, Double-blind Study to Investigate the Safety, Pharmacodynamics, and Preliminary Efficacy of S-606001 as an Add-on to Enzyme Replacement Therapy in Patients With Late-onset Pompe Disease
Brief Title: Study of S-606001 as an Add-on to Enzyme Replacement Therapy (ERT) in Participants With Late-onset Pompe Disease (LOPD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2405N1221; 2025-522146-40 (EudraCT Number)
Record Dates: First submitted 2025-07-25; First posted 2025-08-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pompe Disease
Keywords: Late-onset Pompe disease; Enzyme replacement therapy; LOPD; ERT; S-606001; Muscle glycogen synthase; Liver glycogen synthase; Rare disease; Autosomal disease; Acid alpha-glucosidase; GAA; Glycogen storage disorder; GSD
MeSH Terms: conditions — Glycogen Storage Disease Type II; Rare Diseases; Glycogen Storage Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- S-606001 Low Dose (Experimental): Participants will receive S-606001 at a low dose level twice daily (BID) after a meal for 52 weeks.
  Interventions: Drug: S-606001
- S-606001 High Dose (Experimental): Participants will receive S-606001 at a high dose level BID after a meal for 52 weeks.
  Interventions: Drug: S-606001
- Placebo (Placebo Comparator): Participants will receive S-606001 matching placebo BID after a meal for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-606001 — S-606001 administered orally
  Arms: S-606001 High Dose; S-606001 Low Dose
Drug: Placebo — S-606001 matching placebo administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacodynamics (PD), and exploratory clinical efficacy of S-606001 in adult participants with LOPD as an add-on to ERT.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must be ≥18 years of age and ≥40 kilograms (kg) of body weight at the time of signing the informed consent.
* Participant must have a diagnosis of LOPD based on documentation of 1 of the following:

  1. Deficiency of acid alpha-glucosidase (GAA) enzyme
  2. GAA genotype
* Participant has a %FVC ≥30% and ≤80% in an upright position without mechanical ventilation at screening; or Participant has ≥10% %FVC drop from upright position to supine position and %FVC ≥20% in a supine position.
* Participant performs the 6MWT at screening, as determined by the clinical evaluator, and meets all of the following criteria:

  1. Screening values of 6-minute walk distance (6MWD) are ≥75 meters
  2. Screening values of 6MWD are ≤90% of the predicted value for healthy adults
* Participants must be ERT-experienced, defined as currently receiving ERT and having been receiving ERT for ≥24 months, with no regimen change in the last 6 months.

Key Exclusion Criteria:

* Has a medical condition or any other extenuating circumstance that may pose an undue safety risk to the participant or may compromise his/her ability to comply with or adversely impact protocol requirements.
* Has active infections at screening.
* Malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Current or chronic history of liver disease.
* Known biallelic loss of function mutations whether in glycogenin gene (GYG) or in glycogen phosphorylase muscle associated gene(PYGM) .
* Has received any investigational therapy or pharmacological treatment for Pompe disease, within 30 days or 5 half-lives of the therapy or treatment, whichever is longer, before day 1 or is anticipated to do so during the study.
* Has received gene therapy or small interfering ribonucleic acid (RNA) therapy for Pompe disease.
* Participant, if female, is pregnant or breastfeeding at screening.
* Participant, whether male or female, is planning to conceive a child during the study.

Note: Other protocol-specified inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2027-08-08 (Estimated); Study Completion 2027-08-08 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Percent Forced Vital Capacity (%FVC) at Week 52 | Baseline, Week 52

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Baseline up to Week 53
Plasma Concentration of S-606001 | Up to Week 12
Change From Baseline in Serum Creatine Kinase Levels at Week 52 | Baseline, Week 52
Change From Baseline in 6-minute Walk Test (6MWT) at Week 52 | Baseline, Week 52
Change From Baseline in Pulmonary Function Parameter: Maximal Inspiratory Pressure (MIP) at Week 52 | Baseline, Week 52
Change From Baseline in Pulmonary Function Parameter: Maximal Expiratory Pressure (MEP) at Week 52 | Baseline, Week 52
Change From Baseline in Motor Function Parameter: Gait, Stair, Gower's Maneuver, Chair (GSGC) Score at Week 52 | Baseline, Week 52
Change From Baseline in Patient-Reported Outcomes Measurement Information System Fatigue Short Form 8a (PROMIS-Fatigue-8a) Score at Week 52 | Baseline, Week 52
Change From Baseline in Patient-Reported Outcomes Measurement Information System Physical Function 20-item short form (PROMIS-PF-20) Score at Week 52 | Baseline, Week 52
Change From Baseline in Patient-Reported Outcomes Measurement Information System v2.0 Pain Intensity 3a (PROMIS v2.0 PAIN) Score at Week 52 | Baseline, Week 52
Change From Baseline in 36-item Short Form Health Survey (SF-36) Score at Week 52 | Baseline, Week 52
Change From Baseline in Patient Global Impression of Severity (PGI-S) Score at Week 52 | Baseline, Week 52

CONTACTS AND LOCATIONS:
Locations (28):
- United States (9):
  - University of California - Irvine Medical Center, Irvine, California
  - University of Florida (UF) - Gainesville, Gainesville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Lysosomal and Rare Disorders Research and Treatment Center (LDRTC), Fairfax, Virginia
- UZ Leuven, Leuven, Belgium
- Aarhus University Hospital, Aarhus, Denmark
- France (4):
  - HCL Hopital Pierre Wertheimer, Bron
  - AP-HP Hopital Raymond Poincare, Garches
  - Centre de Reference des Maladies Neuromusculaires et de la SLA - AP-HM Hopital de La Timone, Marseille
  - CHU de Nice - Hopital Pasteur 2 - Centre de reference des Maladies Neuromusculaires, Nice
- Germany (3):
  - Universitaetsklinikum Halle (Saale), Halle
  - SphinCS GmbH, Höchheim
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München
- Italy (2):
  - A.O.U. Policlinico "G. Martino", Messina
  - AOU Citta della Salute e della Scienza di Torino - Ospedale le Molinette, Torino
- Erasmus MC, GE Rotterdam, GE Rotterdam, Netherlands
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (5):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - National Hospital for Neurology & Neurosurgery, London
  - Royal Free London NHS Foundation Trust, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Salford Royal Hospital, Salford